CLINICAL TRIAL: NCT00032630
Title: CSP #517 - Outcomes Following Myocardial Revascularization: On and Off Cardiopulmonary Bypass
Brief Title: Outcomes Following Myocardial Revascularization: On and Off Cardiopulmonary Bypass
Acronym: ROOBY
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 517
Record Dates: First submitted 2002-03-27; First posted 2002-03-28 (Estimated); Results first posted 2014-01-10 (Estimated); Last update posted 2014-05-05 (Estimated); Status verified 2014-04

CONDITIONS: Ischemic Heart Disease
MeSH Terms: conditions — Myocardial Ischemia | interventions — Coronary Artery Bypass, Off-Pump

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1 (Other): Coronary artery bypass - on-pump
  Interventions: Procedure: Coronary artery bypass - on-pump
- Arm 2 (Other): Coronary artery bypass - off-pump
  Interventions: Procedure: Coronary artery bypass - off-pump

INTERVENTIONS:
Procedure: Coronary artery bypass - on-pump — CABG procedure performed on heart lung machine
  Arms: Arm 1
Procedure: Coronary artery bypass - off-pump — CABG procedure performed without the use of the heart lung machine
  Arms: Arm 2

SUMMARY:
Ischemic heart disease is one of the most frequent diagnoses in the VA system. Moreover, 5,819 coronary artery bypass graft (CABG-only) procedures were performed in the VA in Fiscal Year (FY) 1999. Throughout VA and non-VA cardiac surgery programs nationwide, myocardial revascularization is now being performed using two surgical techniques. One technique is performed with cardiopulmonary bypass (CPB) usually with cardioplegic arrest ("on-pump") and the other without CPB on a beating heart ("off-pump"). The overall purpose of this proposed randomized, controlled, clinical trial is to rigorously evaluate the impact of using an on-pump versus off-pump surgical technique for coronary artery bypass graft (CABG-only) procedures (performed with a traditional median sternotomy incision) upon patient clinical outcomes and resource utilization.

DETAILED DESCRIPTION:
Primary Hypotheses: The study has two primary hypotheses to evaluate the impact of using an off-pump versus an on-pump surgical technique for CABG procedures. One is a short term objective to assess the immediate impact of the two surgical techniques while the second assesses the long-term impact of the two techniques: 1) Short-Term Null Hypothesis: For patients having CABG-only procedures performed, there will be no difference in the short-term composite clinical outcome (30 day death or major morbidity) between patients randomized to the on-pump and off-pump procedures, 2) Long-Term Null Hypothesis: For patients undergoing CABG-only procedures, there will be no difference in long-term clinical outcome as measured by one year mortality and/or acute myocardial infarction prior to one year and/or a subsequent revascularization procedure within one year between patients randomized to the on-pump and off-pump procedures.

Secondary Hypotheses: Major secondary objectives are to determine if there are differences in patients undergoing CABG-only procedures using the on-pump and off-pump techniques for 1) long-term completeness of revascularization, 2) one year graft patency and stenosis rates as determined by angiography at one year, and 3) short-term completeness of revascularization. Other secondary objectives are to evaluate the two surgical techniques on 1) changes in neuropsychological function, 2) traditional clinical outcomes, 3) general and disease specific quality of life, and 4) use of system resources.

Intervention: Patients requiring an elective or urgent CABG-only (no other procedures to be done) surgical procedure will be randomized to either the off-pump procedure or to the on-pump procedure.

Primary Outcomes: The short-term primary outcome measure is a composite measure of death, repeat cardiac surgery, new technical support, cardiac arrest, coma, prolonged stroke and/or renal failure requiring dialyses occurring within 30 days of surgery or prior to discharge, whichever is latest. The long-term primary outcome measure is a composite of death, acute myocardial infarction, and/or subsequent revascularization procedure prior to one year post-surgery.

Study Abstract: Ischemic heart disease is one of the most frequent diagnoses in the VA system. Moreover, 5,819 coronary artery bypass graft (CABG-only) procedures were performed in the VA in FY 1999. Throughout VA and non-VA cardiac surgery programs nationwide, myocardial revascularization is now being performed using two surgical techniques. One technique is performed with cardiopulmonary bypass (CPB) usually with cardioplegic arrest ("on-pump") and the other without CPB on a beating heart ("off-pump"). The overall purpose of this proposed randomized, controlled, clinical trial is to rigorously evaluate the impact of using an on-pump versus off-pump surgical technique for coronary artery bypass graft (CABG-only) procedures (performed with a traditional median sternotomy incision) upon patient clinical outcomes and resource utilization.

ELIGIBILITY:
Inclusion Criteria:

* Elective or Urgent CABG
* CABG only procedure to be performed

Exclusion Criteria:

* Patient's surgeon is not a participant that meets study off-pup criteria
* Valve or Valve/CABG procedure
* Emergent, hemodynamically unstable, or in cardiogenic shock preoperatively
* Moderate, moderate, to severe, or severe valvular disease
* Enrolled in another therapeutic or interventional study
* Majority of diffusely diseased distal vessels
* Clinical Care Team has reservations
* History of on-compliance
* Patient preference for treatment arm
* Inability to provide informed consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2203 (Actual)
Dates: Start 2002-04; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frederick Grover, MD, Study Chair — VA Eastern Colorado Health Care System, Denver
Locations (17):
- United States (17):
  - VA Palo Alto Health Care System, Palo Alto, California
  - VA Medical Center, San Francisco, San Francisco, California
  - VA Greater Los Angeles HCS, Sepulveda, Sepulveda, California
  - VA Eastern Colorado Health Care System, Denver, Denver, Colorado
  - VA Medical Center, DC, Washington D.C., District of Columbia
  - North Florida/South Georgia Veterans Health System, Gainesville, Florida
  - VA Medical Center, Miami, Miami, Florida
  - James A. Haley Veterans Hospital, Tampa, Tampa, Florida
  - New Mexico VA Health Care System, Albuquerque, Albuquerque, New Mexico
  - VA Medical Center, Asheville, Asheville, North Carolina
  - VA Medical Center, Durham, Durham, North Carolina
  - VA Medical Center, Cleveland, Cleveland, Ohio
  - VA Medical Center, Portland, Portland, Oregon
  - VA Pittsburgh Health Care System, Pittsburgh, Pennsylvania
  - VA North Texas Health Care System, Dallas, Dallas, Texas
  - VA South Texas Health Care System, San Antonio, San Antonio, Texas
  - Zablocki VA Medical Center, Milwaukee, Milwaukee, Wisconsin

REFERENCES:
- [Result] Shroyer AL, Grover FL, Hattler B, Collins JF, McDonald GO, Kozora E, Lucke JC, Baltz JH, Novitzky D; Veterans Affairs Randomized On/Off Bypass (ROOBY) Study Group. On-pump versus off-pump coronary-artery bypass surgery. N Engl J Med. 2009 Nov 5;361(19):1827-37. doi: 10.1056/NEJMoa0902905. PMID 19890125
- [Result] Wagner TH, Hattler B, Bishawi M, Baltz JH, Collins JF, Quin JA, Grover FL, Shroyer AL; VA #517 Randomized On/Off Bypass (ROOBY) Study Group. On-pump versus off-pump coronary artery bypass surgery: cost-effectiveness analysis alongside a multisite trial. Ann Thorac Surg. 2013 Sep;96(3):770-7. doi: 10.1016/j.athoracsur.2013.04.074. Epub 2013 Aug 2. PMID 23916805
- [Derived] Hattler B, Carr BM, Messenger J, Spertus J, Ebrahimi R, Bishawi M, Quin JA, Almassi GH, Collins JF, Kozora E, Grover FL, Shroyer ALW. Clinical and Angiographic Predictors of Patient-Reported Angina 1 Year After Coronary Artery Bypass Graft Surgery. Circ Cardiovasc Qual Outcomes. 2019 Apr;12(4):e005119. doi: 10.1161/CIRCOUTCOMES.118.005119. PMID 31001997
- [Derived] Bishawi M, Hattler B, Almassi GH, Spertus JA, Quin JA, Collins JF, Grover FL, Shroyer AL; VA #517 Randomized On/Off Bypass (ROOBY) Study Group. Preoperative factors associated with worsening in health-related quality of life following coronary artery bypass grafting in the Randomized On/Off Bypass (ROOBY) trial. Am Heart J. 2018 Apr;198:33-38. doi: 10.1016/j.ahj.2017.12.014. Epub 2017 Dec 24. PMID 29653645
- [Derived] Almassi GH, Carr BM, Bishawi M, Shroyer AL, Quin JA, Hattler B, Wagner TH, Collins JF, Ravichandran P, Cleveland JC, Grover FL, Bakaeen FG; Veterans Affairs #517 Randomized On/Off Bypass (ROOBY) Study Group. Resident versus attending surgeon graft patency and clinical outcomes in on- versus off-pump coronary artery bypass surgery. J Thorac Cardiovasc Surg. 2015 Dec;150(6):1428-35, 1437.e1; discussion 1435-7. doi: 10.1016/j.jtcvs.2015.08.124. Epub 2015 Sep 18. PMID 26470910
- [Derived] Almassi GH, Wagner TH, Carr B, Hattler B, Collins JF, Quin JA, Ebrahimi R, Grover FL, Bishawi M, Shroyer AL; VA #517 Randomized On/Off Bypass (ROOBY) Study Group. Postoperative atrial fibrillation impacts on costs and one-year clinical outcomes: the Veterans Affairs Randomized On/Off Bypass Trial. Ann Thorac Surg. 2015 Jan;99(1):109-14. doi: 10.1016/j.athoracsur.2014.07.035. Epub 2014 Nov 6. PMID 25442992
- [Derived] Hattler B, Messenger JC, Shroyer AL, Collins JF, Haugen SJ, Garcia JA, Baltz JH, Cleveland JC Jr, Novitzky D, Grover FL; Veterans Affairs Randomized On/Off Bypass (ROOBY) Study Group. Off-Pump coronary artery bypass surgery is associated with worse arterial and saphenous vein graft patency and less effective revascularization: Results from the Veterans Affairs Randomized On/Off Bypass (ROOBY) trial. Circulation. 2012 Jun 12;125(23):2827-35. doi: 10.1161/CIRCULATIONAHA.111.069260. Epub 2012 May 16. PMID 22592900
- [Derived] Novitzky D, Baltz JH, Hattler B, Collins JF, Kozora E, Shroyer AL, Grover FL. Outcomes after conversion in the Veterans Affairs randomized on versus off bypass trial. Ann Thorac Surg. 2011 Dec;92(6):2147-54. doi: 10.1016/j.athoracsur.2011.05.122. Epub 2011 Oct 5. PMID 21978872
- [Derived] Zenati MA, Shroyer AL, Collins JF, Hattler B, Ota T, Almassi GH, Amidi M, Novitzky D, Grover FL, Sonel AF. Impact of endoscopic versus open saphenous vein harvest technique on late coronary artery bypass grafting patient outcomes in the ROOBY (Randomized On/Off Bypass) Trial. J Thorac Cardiovasc Surg. 2011 Feb;141(2):338-44. doi: 10.1016/j.jtcvs.2010.10.004. Epub 2010 Dec 3. PMID 21130476

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From February 2002 to May 2007, a total of 9663 patients who were scheduled for urgent or elective Coronary Artery Bypass Graft (CABG) were screened for enrollment. Of these, 7460 patients were excluded, mostly because of diffusely diseased or small coronary arteries. Overall,1099 patients were randomized to on-pump and 1104 randomized to off-pump
Groups:
- On Pump: Coronary artery bypass performed on a non beating heart using a heart-lung machine
- Off Pump: Coronary artery bypass performed on a beating heart with no heart-lung machine
Period: Overall Study
Arm/Group | On Pump | Off Pump
Started | 1099 | 1104
Completed | 1050 | 1061
Not Completed | 49 | 43

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | On Pump | Off Pump | Total
Number analyzed (Participants) | 1099 | 1104 | 2203
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 699 | 671 | 1370
  >=65 years | 400 | 433 | 833
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.5 (8.5) | 63.0 (8.5) | 62.74 (8.49)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 7 | 13
  Male | 1093 | 1097 | 2190
Region of Enrollment [Number; unit: participants]
  United States | 1099 | 1104 | 2203

OUTCOME MEASURES:

1. Primary Outcome: Short-term End Point
Description: Short-term end point was a composite of death or major complications (reoperation, new mechanical support, cardiac arrest, coma, stroke, or renal failure requiring dialysis) occuring within 30 days after surgery or before discharge, whichever was later.
Time Frame: 30 day
Measure: Number; unit: participants
Arm/Group | On Pump | Off Pump
Number analyzed (Participants) | 1099 | 1104
participants | 61 [0.1 to 4.9] | 77 [0.1 to 4.9]

2. Primary Outcome: Long-term Composite
Description: Long-term composite endpoint was death from any cause within 1 year, nonfatal myocardial infarction between 30 days and 1 year, or repeat revascularization between 30 days and 1 year.
Time Frame: one-year
Measure: Number; unit: Participants
Arm/Group | On Pump | Off Pump
Number analyzed (Participants) | 1050 | 1061
Participants | 78 | 105

ADVERSE EVENTS:
Arm/Group | On Pump | Off Pump
Serious Adverse Events (participants affected / at risk) | 201/1099 | 220/1104
Other Adverse Events (participants affected / at risk) | 0/1099 | 0/1104
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | On Pump (N=1099) | Off Pump (N=1104)
Chest Pain (Cardiac disorders) | 64 (64) | 69 (69)
Congestive Heart Failure (Cardiac disorders) | 33 (33) | 30 (30)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 32 (32) | 30 (30)
Myocardial Infarction (Cardiac disorders) | 18 (18) | 36 (36)
CVA (Nervous system disorders) | 19 (19) | 19 (19)
Atrial Fibrillation (Cardiac disorders) | 15 (15) | 22 (22)
Wound Infection (Infections and infestations) | 20 (20) | 14 (14)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes